CLINICAL TRIAL: NCT02389933
Title: Multiple Patient Program to Ensure Access to LCZ696 Treatment to Patients Diagnosed With Heart Failure With Reduced Ejection Fraction (HF-rEF)
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696B2318M
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HF-rEF)
Keywords: Multiple Patient Program, LCZ696, heart failure, heart failure with reduced ejection fraction, HF-rEF
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: LCZ696 — immediate release film coated tablet in 50 mg, 100 mg, 200 mg, and 400 mg strengths for oral administration.

SUMMARY:
Novartis has set up this global Multiple Patient Program (MPP) treatment plan to provide access to life-saving treatment with LCZ696 for patients that were not previously exposed to LCZ696 but have no other option to receive LCZ696 in their country prior to market authorization OR commercial availability, based on local regulatory and legal requirements.

ELIGIBILITY:
Inclusion criteria

The patient(s) for whom the MPP is sought meets all of the following:

* Is suffering from a serious or life-threatening disease or condition
* Does not have access to a comparable or satisfactory alternative treatment (i.e., comparable or satisfactory treatment is not available or does not exist)
* Patient should be on optimized standard of care treatment, including treatment with ARBs or ACEI, beta-blockers and MRA;
* Intolerance to evidence-based target doses should be documented by the treating physician
* Meets any other relevant medical criteria for compassionate use of the investigational product

Patients eligible for inclusion in this program have to fulfill all of the following criteria:

1. Adult patients (but not younger than 18 year old) will be included, upon completion of written informed consent before any assessment is performed.
2. Patients with a diagnosis of CHF NYHA class II-IV and reduced ejection fraction:

   • LVEF ≤ 35% at the time of screening for participation in the program (any local measurement, made within the past 6 months using echocardiography, MUGA, CT scanning, MRI or ventricular angiography is acceptable, provided there are no subsequent measurement above 35%)
3. Patient had a hospitalization for HF within the last 12 months
4. Patients must be on an ACEI or an ARB at a stable dose for at least 4 weeks prior to starting treatment with LCZ696
5. Patients must be treated with a β-blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks prior to starting treatment with LCZ696 (reason should be documented for patients not on CHF target doses per local guidelines, or in absence of that medication).
6. An aldosterone antagonist should also be considered in all patients, taking account of renal function, serum potassium and tolerability. If given, the dose of aldosterone antagonist should be optimized according to guideline recommendations and patient tolerability, and should be stable for at least 4 weeks prior to starting treatment with LCZ696

Exclusion criteria

Patients fulfilling any of the following criteria are not eligible for inclusion in this program:

1. The patient is eligible for participation in any of the IMP's ongoing clinical trials
2. The patient has recently completed a clinical trial that has been terminated and other options (e.g., trial extensions, amendments, etc.) are available to continue a similar treatment.
3. The patient is being transferred from an ongoing clinical trial for which the patient is still eligible for participation
4. History of hypersensitivity or allergy to LCZ696 or to any of its metabolites; to drugs of similar chemical classes, ARBs, or NEP inhibitors; as well as known or suspected contraindications to LCZ696
5. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
6. Previous history of intolerance to recommended target doses of ARBs
7. Known history of angioedema
8. Requirement of concomitant treatment with both ACEIs and ARBs
9. Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy)
10. Symptomatic hypotension and/or a SBP less than 100 mm Hg over the last 4 weeks prior to starting treatment with LCZ696
11. Estimated GFR below 30 mL/min/1.73m2 as measured by the simplified MDRD formula
12. Presence of bilateral renal artery stenosis
13. Serum potassium above 5.2 mmol/L during the week prior to starting treatment with LCZ696
14. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major CV surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within the 3 months prior to starting treatment with LCZ696
15. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after the schedule date to start treatment with LCZ696
16. Implantation of a cardiac resynchronization therapy pacemaker (CRT-P) or a cardiac resynchronization therapy defibrillator (CRT-D) or upgrading of an existing conventional pacemaker or an implantable cardioverter defibrillator (ICD) to CRT device within 3 months prior to starting treatment with LCZ696, or intent to implant such a device.

    Also, patients who had implantation of a conventional pacemaker or an ICD or had a revision of a pacemaker or other device leads within 1 month before starting treatment with LCZ696 are excluded.
17. Heart transplant or ventricular assistance device (VAD) or intent to transplant (on transplant list) or implant a VAD
18. History of severe pulmonary disease
19. Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to starting treatment with LCZ696
20. Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months prior to starting treatment with LCZ696
21. Symptomatic bradycardia or second or third degree heart block without a pacemaker
22. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation
23. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis
24. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs, including but not limited to any of the following:

    * History of active inflammatory bowel disease during the 12 months before starting treatment with LCZ696.
    * Current duodenal or gastric ulcers during the 3 months prior to starting treatment with LCZ696
    * Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x ULN prior to starting treatment with LCZ696, history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt
    * Active treatment with cholestyramine or colestipol resins
25. Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 3 x ULN prior to starting treatment with LCZ696, history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt
26. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (above 5 mIU/mL)
27. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method (if accepted by the local regulatory authority and ethics committee) or a barrier method plus a hormonal method

    * Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progesterone agent.
    * Reliable contraception should be maintained throughout the treatment and for 7 days after LCZ696 treatment discontinuation
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea, or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
28. Presence of any other disease with a life expectancy of < 3 years
29. Any condition, not identified in the protocol that in the opinion of the treating physician is likely to prevent the patient from safely tolerating LCZ696 or complying with the requirements of the therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (220):
- Novartis Investigative Site, Vero Beach, Florida, United States
- Australia (3):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, North Ryde, New South Wales
  - Novartis Investigative Site, Perth, Western Australia
- Austria (4):
  - Novartis Investigative Site, Krems
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Sankt Pölten
  - Novartis Investigative Site, Vienna
- Brazil (4):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
- Novartis Investigative Site, Varaždin, HRV, Croatia
- Cyprus (2):
  - Novartis Investigative Site, Limassol
  - Novartis Investigative Site, Nicosia
- France (78):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Bron, Cedex
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Saint-Denis, France / La Reunion
  - Novartis Investigative Site, Brest Armees, France
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Amilly
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Antibes
  - Novartis Investigative Site, Aressy
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayeux
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Cambrai
  - Novartis Investigative Site, Cannes
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Chaumont
  - Novartis Investigative Site, Cherbourg Octeville
  - Novartis Investigative Site, Clamart
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Contamine-sur-Arve
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Cornebarrieu
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Eaubonne
  - Novartis Investigative Site, Honfleur
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, La Tronche
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Mâcon
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Metz-Tessy
  - Novartis Investigative Site, Monaco
  - Novartis Investigative Site, Montbéliard
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Morlaix
  - Novartis Investigative Site, Moulins
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Neuilly-sur-Seine
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pau
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Pont-l'Abbé
  - Novartis Investigative Site, Pontarlier
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Rumilly
  - Novartis Investigative Site, Saint-Denis
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Saint-Germain-en-Laye
  - Novartis Investigative Site, Saint-Palais
  - Novartis Investigative Site, St.-Jean
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Thonon-les-Bains
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Valenciennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Vichy
  - Novartis Investigative Site, Villefranche-sur-Saône
  - Novartis Investigative Site, Wattrelos
- Germany (53):
  - Novartis Investigative Site, Süderholz, OT Bartmannshagen
  - Novartis Investigative Site, Ahlen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Endbach
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Kreuznach
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Diepholz
  - Novartis Investigative Site, Dinslaken
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eilenburg
  - Novartis Investigative Site, Eschwege
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Friedrichroda
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Gronau
  - Novartis Investigative Site, Günzburg
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Haßfurt
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Hohenstein-Ernstthal
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Köthen
  - Novartis Investigative Site, Lauchringen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marl
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Pressath
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Wildeshausen
  - Novartis Investigative Site, Wolfratshausen
  - Novartis Investigative Site, Würzburg
- Greece (29):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Heraklion - Crete, Greece
  - Novartis Investigative Site, Thesaloniki, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Tripoli, GR
  - Novartis Investigative Site, Voula, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Chios
  - Novartis Investigative Site, Corfu
  - Novartis Investigative Site, Edessa
  - Novartis Investigative Site, Elefsina
  - Novartis Investigative Site, Glyfada
  - Novartis Investigative Site, Heraklion
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Kalamata
  - Novartis Investigative Site, Karditsa
  - Novartis Investigative Site, Katerini
  - Novartis Investigative Site, Kavala
  - Novartis Investigative Site, Kilkis
  - Novartis Investigative Site, Kozani
  - Novartis Investigative Site, Marousi
  - Novartis Investigative Site, Piraeus
  - Novartis Investigative Site, Rio Patra
  - Novartis Investigative Site, Thessaloniki
  - Novartis Investigative Site, Volos
- Ireland (2):
  - Novartis Investigative Site, Co Dublin, Ireland
  - Novartis Investigative Site, Dublin
- Lebanon (4):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
  - Novartis Investigative Site, Tripoli
- Novartis Investigative Site, Msida, Malta
- Novartis Investigative Site, Panama City, Panama
- Philippines (3):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Manila
- Novartis Investigative Site, Ljubljana, Slovenia
- Spain (30):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Garanada, Andalusia
  - Novartis Investigative Site, Jerez de la Frontera, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Utrera, Andalusia
  - Novartis Investigative Site, Baleares, Balearic Islands
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Galdakano, Basque Country
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Torrelavega, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Salt, Catalonia
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Pontevedra, Galicia
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, Marbella, Malaga
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, El Palmar (Murcia)
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Zaragoza
- Novartis Investigative Site, Lucerne, Canton of Lucerne, Switzerland
- United Arab Emirates (2):
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Ras al-Khaimah